CLINICAL TRIAL: NCT06968962
Title: A Multicenter, Randomized, Controlled, Double-blind, and Non-inferiority Clinical Trial to Compare the Efficacy of Sequential to Initial Combination Therapy in Patients With Pulmonary Arterial Hypertension
Brief Title: Comparison of Sequential to Initial Combination Therapy in PAH
Acronym: ORIENTATION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Huzhou Central Hospital (Other); Ningbo Medical Center Lihuili Hospital (Other Government); First Affiliated Hospital of Ningbo University (Network); Ningbo No.2 Hospital (Other); Affiliated Hospital of Jiaxing University (Other); The Second Affiliated Hospital of Jiaxing University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Shanghai Pulmonary Hospital affiliated to Tongji University (Unknown); Taizhou Hospital (Other); Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, JianAn Wang, Professor, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YAN2024-1201
Record Dates: First submitted 2025-04-20; First posted 2025-05-13 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Arterial Hypertension (PAH)
Keywords: Sequential combination therapy; Initial combination therapy; Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Tadalafil; ambrisentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Initial combination therapy (Active Comparator): Patients will receive dual combination therapy with Ambrisentan and Tadalafil immediately after randomization.
  Interventions: Drug: Tadalafil; Drug: Ambrisentan
- Sequential combination therapy (B1 group) (Experimental): Patients will receive Ambrisentan and Tadalafil mimic first, with sequential addition of Tadalafil if low risk status was not achived at month 4, or 8, or 12.
  Interventions: Drug: Ambrisentan; Drug: Tadalafil mimic
- Sequential combination therapy (B2 group) (Experimental): Patients will receive Tadalafil and Ambrisentan mimic first, with sequential addition of Ambrisentan if low risk status was not achived at month 4, or 8, or 12.
  Interventions: Drug: Tadalafil; Drug: Ambrisentan mimic

INTERVENTIONS:
Drug: Tadalafil — Target dose 40 mg OD
  Arms: Initial combination therapy; Sequential combination therapy (B2 group)
Drug: Ambrisentan — Target dose 10 mg OD
  Arms: Initial combination therapy; Sequential combination therapy (B1 group)
Drug: Ambrisentan mimic — Ambrisentan mimic will switch to Ambrisentan if low risk status was not achived at month 4, or 8, or 12.
  Arms: Sequential combination therapy (B2 group)
Drug: Tadalafil mimic — Tadalafil mimic will switch to Tadalafil if low risk status was not achived at month 4, or 8, or 12.
  Arms: Sequential combination therapy (B1 group)

SUMMARY:
This is a multicenter, randomized, controlled, double-blind, and non-inferiority clinical trial to compare the efficacy of sequential to initial combination therapy in patients with pulmonary arterial hypertension (PAH). Ambrisentan and Tadalafil will be used in the study. Our research hypothesis is that the efficacy of sequential combination therapy in PAH patients is not inferior to the initial combination therapy as the primary efficacy endpoint is the change in 6MWD at month 12 from baseline.

DETAILED DESCRIPTION:
This is a multicenter, randomized, controlled, double-blind, and non-inferiority clinical trial to compare the efficacy of sequential to initial combination therapy in symptomatic patients with PAH (WHO functional class I-III) and assessed as low-risk or moderate-risk based on 2022 ESC/ERS risk stratification. Subjects must not have previously received chronic PAH therapy (i.e., prostanoids, ERAs, or PDE-5 inhibitors) within 4 weeks prior to Screening.

Treatment Escalation

1. The investigators will conduct a risk stratification assessment based on COMPERA 2.0 every 4 months, i.e. at month 4, 8, and 12.

2. If the patient meets the low-risk criteria, their current treatment regimen will be maintained, and both the patient and the investigator will be unaware of the specific regimen.

3. If the patient does not meet the low-risk criteria:

1. No clinical failure events have occurred: The first step is to escalate to blinded dual therapy.

   1. The investigator initiates a request for blinded dual therapy, and the pharmacist informs the investigator that the treatment plan has been upgraded as requested.
   2. If the patient is currently on mono therapy, the pharmacist will escalate the regimen to dual therapy.
   3. If the patient is currently in the initial combination therapy group or has already escalated to blinded dual therapy, the pharmacist will maintain the current dual therapy regimen.
2. If any clinical failure event occurs at any time, as determined by the Clinical Event Evaluation Committee:

   1. Escalate to blinded dual therapy as described above
   2. Or add prostacyclin analogue
   3. Or add IP receptor agonist
   4. Or transition of Tadalafil to Riociguat
   5. Or add Sotatercept

Primary efficacy endpoint is exercise capacity, as the change in 6MWD at month 12 from baseline. Secondary efficacy endpoints will include time to clinical failure events during the 12-month treatment period, and others detailed in outcome measures.

Study duration will be approximately 4 years. A non-inferiority test will be conducted based on the mean difference and 95% CI of the change in 6MWD between groups after 12 months of treatment following randomization. An unblinded, external, independent DSMB will monitor participants' data and safety throughout the course of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 80 years and weight ≥ 40 kg.
2. WHO functional classification I-III.
3. Diagnosed with PAH caused or related to the following:

1) Idiopathic PAH 2) Hereditary PAH 3) Associated PAH:

1. Connective tissue diseases (e.g., scleroderma, systemic lupus erythematosus, mixed connective tissue disease, etc.)
2. Drug or toxin exposure
3. Corrected congenital heart diseases for more than 1 year (e.g., atrial septal defect, ventricular septal defect, and patent ductus arteriosus) 4. Risk stratification assessed as low-risk or intermediate-risk according to the 2022 ESC/ERS guidelines.

   5. Right heart catheterization meets the following criteria (end-expiratory data, original waveform must be retained for quality control):

   1) Mean pulmonary artery pressure ≥ 25 mmHg 2) Pulmonary vascular resistance ≥ 3 Wood units 3) Pulmonary artery wedge pressure (PAWP) ≤ 15 mmHg 4) Cardiac output measurement requirements: thermal dilution or direct Fick method; indirect Fick method does not meet study criteria.

   6. Pulmonary function tests meet the following criteria:

   1） Total lung capacity (TLC) ≥ 60% of the predicted normal value; 2） Forced expiratory volume in the first second (FEV1) ≥ 55% of the predicted normal value; 3） DLCO_SB ≥ 40% of the predicted normal value. 7. Baseline 6MWD more than 100 meters repeated twice at screening (measured at least 4 hours apart, but no longer than 1 week), and both values are within 15% of each other (calculated from the highest value) 8. In a resting state, without supplemental oxygen, arterial oxygen saturation (SaO2) ≥ 88%.

   9. No participation in cardiopulmonary rehabilitation training programs within 12 weeks prior to the screening visit.

   10. Females of childbearing potential must agree to use contraception until the end of the study.

   11. No participation in clinical studies involving other investigational drugs or devices throughout the study duration.

   12. Ability to understand the informed consent form and sign it.

   Exclusion Criteria:

   1. Other types of pulmonary arterial hypertension (PAH)
   1. Other types of PAH, such as HIV-related PAH, schistosomiasis-related PAH, etc.
   2. Pulmonary arterial hypertension associated with portal hypertension
   3. Pulmonary vein occlusive disease or pulmonary capillary hemangiomatosis 2. Group 4 PH, e.g. Chronic thromboembolic pulmonary hypertension 3. Group 2 PH, i.e., PH associated with left heart disease 4. Group 3 PH, i.e., PH associated with lung disease or hypoxia 5. Group 5 PH, i.e., PH with unclear mechanisms or multi-mechanism 6. PAH Therapy

   1) Subjects who have received PAH therapy (such as PDE5 inhibitors, ERAs, or chronic prostacyclin therapy) within 4 weeks prior to the screening visit.

   2) Subjects who have ever received ERA therapy (e.g., macitentan) or PDE5 inhibitor therapy (e.g., sildenafil) and discontinued due to tolerance issues unrelated to liver dysfunction.

   3) Subjects known to have an allergy to the investigational product, its metabolites, or excipients.

   7. Other Therapies
   1. Subjects who have received intravenous inotropes (e.g., dobutamine) within 2 weeks prior to the screening visit.
   2. Subjects receiving protease inhibitors, systemic ketoconazole, or systemic itraconazole therapy.
   3. Subjects receiving strong CYP3A4 inducers (e.g., rifampicin).
   4. Subjects who have received unstable doses of calcium channel blockers or HMG-CoA reductase inhibitors (statins) within 4 weeks prior to the screening visit (eligible subjects must not have changed doses within 4 weeks prior to the screening visit).
   5. Subjects with a history of angina or who have received long-acting or short-acting nitrate treatment within the 12 weeks prior to the visit.

   8. Laboratory Tests at Screening

   1） Serum ALT or AST laboratory values > 2 times the upper limit of normal at screening.

   2） Serum bilirubin laboratory values > 1.5 times the upper limit of normal at screening.

   3） Severe renal impairment (estimated glomerular filtration rate < 45 mL/min/1.73m3) at screening.

   9. Medical History/Current Medical Conditions
   1. Severe liver dysfunction (Child-Pugh Class C, with or without cirrhosis) at screening.
   2. Significant anemia in the opinion of the investigator.
   3. History of bleeding disorders or significant active peptic ulcers.
   4. Uncontrolled hypertension (≥ 180/110 mmHg) at screening.
   5. Severe hypotension (< 90/50 mmHg) at screening.
   6. Myocardial infarction within 3 months prior to screening.
   7. Clinically significant aortic or mitral valve disease, constrictive pericarditis, restrictive or congestive cardiomyopathy, life-threatening arrhythmias, significant left ventricular dysfunction, left ventricular outflow tract obstruction, symptomatic coronary artery disease, autonomic hypotension, or circulatory failure.
   8. History of non-arteritic anterior ischemic optic neuropathy.
   9. Hereditary degenerative retinal disease (e.g., retinitis pigmentosa).
   10. Significant fluid retention in the opinion of the investigator.
   11. Subjects with cardiovascular, liver, kidney, hematologic, gastrointestinal, immune, endocrine, metabolic, or central nervous system diseases that the investigator believes may adversely affect the subject's safety and/or the efficacy of the investigational product or significantly impact the subject's lifespan.
   12. History of malignant tumors within the past 5 years, except for those with local, non-metastatic basal cell carcinoma, cervical carcinoma in situ, or prostate cancer who are not anticipated to receive radiotherapy, chemotherapy, and/or surgical interventions or initiate hormonal therapy during the study period.
   13. Pregnant or breastfeeding female subjects.
   14. Subjects with demonstrated poor compliance.
   15. History of alcohol abuse or illicit drug use within 1 year.
   16. Participation in clinical studies involving another investigational drug or device within 4 weeks prior to the screening visit.

   Subjects who fail inclusion/exclusion criteria may be re-screened once.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The change of 6MWD at month 12 from baseline | Baseline and Month 12
  The 6MWD was the distance walked in 6 minutes as a measure of functional capacity. This was assessed using the 6-minute walk test (6MWT).

SECONDARY OUTCOMES:
Time to clinical failure events during the 12-month treatment period. | During the 12-month treatment period
  Definition of Clinical Failure Events:
  1. Death (all-cause)
  2. Hospitalization due to worsening PAH (adjudicated)
     1. Any hospitalization for worsening
     2. PAH Lung or heart/lung transplantation
     3. Atrial septostomy
     4. Initiation of parenteral prostanoid therapy
     5. Need to initiate rescue therapy
     <!-- -->
     1. Switch Tadalafil to Macitentan
     2. Add Selexipag
     3. Add Sotatercept
  3. Disease progression (adjudicated)
     1. Decrease in 6MWD of more than 15% from baseline
     2. Concurrent presence of WHO functional class III or IV symptoms (continuously observed in follow-up after baseline with at least 14 days apart)
  4. Unsatisfactory long-term clinical response (Adjudicated, all criteria must be met)
     1. Receiving at least one dose of randomized treatment and being in the study for at least 6 months
     2. A decrease in 6MWD from baseline in two assessments separated by at least 14 days
     3. WHO functional class III symptoms assessed at two visits separated by > 6 months
Low-risk status achievement rates. | Month 4, 8 and 12
  Risk stratification will be assess according to COMPERA 2.0, which includes WHO functional class, 6MWD, and BNP or NT-proBNP.
The change of NT-proBNP at month 12 from baseline | Baseline and Month 12
  NT-proBNP is a circulating biomarker that reflects cardiac afterload, this will be measured by central lab.
The change of WHO functional class at month 12 from baseline | Baseline and Month 12
  WHO functional classification for PAH ranges from Class I (no limitation in physical activity, no dyspnea with normal activity), Class II (slight limitation of physical activity), Class III (marked limitation of physical activity) and Class IV (cannot perform a physical activity without any symptoms, dyspnea at rest).
The change of pulmonary vascular resistance at month 12 from baseline | Baseline and Month 12
  Pulmonary vascular resistance is a hemodynamic variable of pulmonary circulation and was measured by right heart catheterization.
Percentage of subjects receiving mono, dual or triple therapy | Month 4, 8, and 12
Percentage of subjects with satisfactory clinical response | Month 8, and 12
  1. An increase of 10% in 6MWD compared to baseline.
  2. Improvement or maintenance of WHO class I or II symptoms.
  3. No clinical failure events occurring during the study.
The change of EmPHasis-10 score from baseline | Baseline, Month 4, 8, and 12
  The EmPHasis-10 questionnaire is used during clinical assessments to estimate how pulmonary hypertension affects patients' life (range: 0=no impact to 5=severe impact). A higher score indicated more severe impact.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No